CLINICAL TRIAL: NCT03527628
Title: A Phase II, Multicenter, Open Label Study of Treatment Intensification With ACVD and Brentuximab-Vedotin in Advanced-stage Hodgkin Lymphoma Patients With a Positive Interim PET Scan After 2 ABVD Cycles
Brief Title: OPTmizing Advanced Stage HodgkIn LymphoMa patIentS Therapy
Acronym: (Optimist)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC-16/150
Record Dates: First submitted 2017-12-12; First posted 2018-05-17 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Classical Hodgkin Lymphoma; Hodgkin Lymphoma (Category); Hodgkin Disease; Hodgkin Lymphoma
Keywords: Stage II B Classical Hodgkin Lymphoma; Stage III Classical Hodgkin Lymphoma; Stage IV Classical Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Doxorubicin; Cyclophosphamide; Vinblastine; Dacarbazine; Brentuximab Vedotin; Bleomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with PET-2 Negative Result (Other): After 2 ABVD cycles an interim PET-2 will be performed, and treatment will be adapted according to to PET results
  PET-2 negative patients will be treated with 4 cycles of ACVD (Adriamycin, Cyclophosphamide, Vinblastine And Dacarbazine)
  Interventions: Drug: Adriamycin; Drug: Cyclophosphamide; Drug: Vinblastine; Drug: Dacarbazine; Drug: ABVD
- Patients with PET-2 Positive Result (Other): After 2 ABVD cycles an interim PET-2 will be performed, and treatment will be adapted according to to PET results
  PET-2 positive patients will be treated with 4 cycles of ACVD with addition of Brentuximab Vedotin
  Interventions: Drug: Adriamycin; Drug: Cyclophosphamide; Drug: Vinblastine; Drug: Dacarbazine; Drug: Brentuximab Vedotin; Drug: ABVD

INTERVENTIONS:
Drug: Adriamycin — 25mg/m2 Bolus injection via fast running drip of 0.9% NaCl in days 1 and 15 of each 28 day cycle.
  Other Names: Doxorubicin
Drug: Cyclophosphamide — 400mg/m2 Infusion in 500ml sodium chloride 0.9%over 30min. in days 1 and 15 of each 28 day cycle
  Other Names: Cytoxan®; Neosar®; Cycloblastin; Revimmune
Drug: Vinblastine — 6mg/m2 Intravenous infusion in 50ml sodium chloride 0.9% over 10 minutes, in days 1 and 15 of each 28 day cycle
  Other Names: Velbe ®
Drug: Dacarbazine — 375mg/m2 Infusion in 500mls 0.9% NaCI over least 60mins. in days 1 and 15 of each 28 day cycle
  Other Names: DTIC
Drug: Brentuximab Vedotin — 1.2mg/kg Intravenous infusion, in days 1 and 15 of each 28 day cycle
  Other Names: ADCETRIS®; SGN-35
  Arms: Patients with PET-2 Positive Result
Drug: ABVD — All enrolled patients receive 2 cycles of ABVD (Adriamycin 25mg/m2, Bleomycin10,000units/m2, Vinblastine 6mg/m2 and Dacarbazine 375mg/m2)
  Other Names: (Adriamycin, Bleomycin, Vinblastine and Dacarbazine )

SUMMARY:
This is a prospective, multi-center, open-label, phase II clinical trial, aims to assess the effectiveness of the combination ACVD (Adriamycin, Cyclophosphamide, Vinblastine and Dacarbazine) and BV (Brentuximab Vedotin) in PET-2 positive advanced-stage HL patients, in order to improve the overall long-term disease control in the entire cohort of advanced-stage HL.

DETAILED DESCRIPTION:
With the aim of reducing Blemoycin pulmonary injury (BPI) , Bleomycin was withdrawn and substituted with Cyclophosphamide (ACVD cycle) in patients with a PET-2 negative. All advanced stage HL patients will receive 2 cycles of the standard treatment ABVD and assessed with PET-2 scan.

Knowing that Cyclophosphamide toxicities include cytopenias, amenorrhea and male infertility. These toxicities are mainly dependent on the total cumulative dose. Doses less than 4 g/m2 are not associated with sterility or major toxicity, doses higher than this can lead to azoospermia which was reversible in many cases therefore the cumulative dose will be used in this study is 3200 mg. Additionally, Brentuximab Vedotin has shown significant activity in relapsed refractory HL with minor toxicities.

PET scan after 2 cycles of ABVD has proven to be an excellent tool to identify patients that will have long term PFS of 95% when it is negative and only progression-free survival (PFS) of less than 15% when it is positive.

The primary endpoint of the study will be to assess the overall 3-Y PFS of the entire cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* All the following parameters should be met

  * Newly diagnosed untreated ,histologically proven CD30 positive classical Hodgkin Lymphoma (cHL)
  * Advanced stage (Stage IIB to IVB) as defined by Ann Arbor Staging System (Appendix 1)
  * Age ≥ 14, < 60 years
  * ECOG performance status 0-2
  * Written informed consent for the trial
  * Adequate contraceptive precautions for all patients of childbearing potential
  * All prognostic group

Exclusion Criteria:

* Any of the following:

  * Pregnant or lactating women.
  * Presence of the following:

    1. Heart failure with LVEF <50%
    2. Liver enzymes, >2 ULN not attributed to Hodgkin Lymphoma.
    3. Another malignancy that is currently clinically significant or requires active intervention
  * Early-stage disease (Stage I- IIA).
  * Patients who are already participating to another clinical trial.
  * Known history of HIV seropositive status
  * ECOG performance status 3-4
  * Creatinin clearance <50 ml/min
  * Prior treatment for Hodgkin Lymphoma excluding steroids
  * Medical or psychiatric conditions compromising the patient's ability to give informed consent
  * Patients with serious active infection
  * Pre-existing peripheral neuropathy (grade 2 or more).

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 220 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-01-15 (Estimated); Study Completion 2022-01-15 (Estimated)

PRIMARY OUTCOMES:
]Progression Free Survival (PFS) | 3 years
  PFS is estimated from the date of diagnosis until the date of first disease progression or relapse, death for any cause.
  Superior overall 3 year progression-free survival of patients with PET 2 positive after 2 cycles of ABVD with ACVD and BV compared to historical control of ABVD treated patients and PET 2 negative patients with ACVD only after 2 cycles of ABVD.

SECONDARY OUTCOMES:
Overall Survival (OS) | 5 years
  Superior overall survival of PET 2 positive patients treated with ACVD + BV after 2 cycles of ABVD and PET 2 negative treated with ACVD after 2 cycles of ABVD. It is estimated from the date of diagnosis up to study completion or death, whichever came first, assessed up to 5 years.

OTHER OUTCOMES:
Reduction of lung toxicity | 6 months
  The ability of ACVD to reduce lung toxicity as compared to ABVD by performing a pulmonary function test (PFT) at baseline and end of treatment
Overall toxicity | 6 months
  The feasibility of the entire program in terms of grade 3 or 4 NCICTCAE or WHO toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Hejazi, MD, Principal Investigator — King Abdulaziz Medical City, Ministry of National Gaurd (KAMC)
Locations (1):
- King Abdulaziz Medical City, Ministry of National Guard, Riyadh, Saudi Arabia